CLINICAL TRIAL: NCT01036633
Title: Use of an Infrared Thermometer to Grade the Severity of Oral Mucositis in Patients Undergoing Antineoplastic Chemotherapy
Brief Title: Oral Mucositis in Patients Undergoing Antineoplastic Chemotherapy
Acronym: Mucositis
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 110227
Record Dates: First submitted 2009-10-08; First posted 2009-12-21 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Oral Mucositis
Keywords: mucositis
MeSH Terms: conditions — Stomatitis; Mucositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group no mucositis: Control patients with multiple myeloma who are not currently receiving chemotherapy and who do not suffer from oral mucositis
  Interventions: Device: Infrared Thermometer
- Non-control Group Mucositis: Patients with multiple myeloma suffering from WHO Grade 3/4 Oral Mucositis
  Interventions: Device: Infrared Thermometer

INTERVENTIONS:
Device: Infrared Thermometer — The infrared thermometer will be used to grade the severity of oral mucositis in patients undergoing antineoplastic chemotherapy for multiple myeloma. The photothermal camera will be used to take intraoral digital images of the mouth.

SUMMARY:
The purpose of this study was to:

1. To investigate the feasibility of using infrared (IR) thermometer to grade the severity of oral mucositis in patients with multiple myeloma undergoing chemotherapy.
2. To obtain preliminary data on the most optimal method of scoring the severity of oral mucositis by comparing the results obtained using the IR thermometer to the World Health Organization (WHO) mucositis grading system and the patient self-assessment questionnaire.
3. To Investigate the correlation between the quantitative readings obtained from oral mucosa with the IR thermometer.

DETAILED DESCRIPTION:
Several grading systems for oral mucositis are available including those of the World Health Organization (WHO), Radiation Therapy Oncology Group (RTOG), Western Consortium for Cancer Nursing Research WCCNR, and the National Cancer Institute Common Toxicity Criteria (NCICTC) and others However, all of these oral mucositis grading systems rely on visual examination and are therefore subjective and operator-dependent tools and suffer from significant interpersonal variability (6). With the current improvements in medicine and technology, there is definitely a need for a more objective, easy to perform, non-invasive, affordable, quantitative and reproducible tool that is operator-independent to assess the severity of oral mucositis. The introduction of such a tool would greatly improve our ability to compare the oral mucosal toxicity of antineoplastic therapies and the efficacy of various mucoprotective therapies. Furthermore, the use of such a tool can be extended to patients undergoing radiation treatment with or without chemotherapy for various malignancies including head and neck cancers.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma receiving chemotherapy Grade 3/4 Mucositis

Exclusion Criteria:

* Women of child bearing potential who are unable to take adequate contraceptive precautions, have + pregnancy test w/in 24 hrs prior to study, pregnant, currently breastfeeding will not be able to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving Chemotherapy for Multiple Myeloma and suffering with mucositis
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To investigate the feasibility of using an infrared (IR) thermometer to grade the severity of oral mucositis in patients with multiple myeloma undergoing chemotherapy | 24 months

SECONDARY OUTCOMES:
Investigating the correlation between the quantitative readings obtained from oral mucosa with an IR thermometer. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Emre Vural, MD, Principal Investigator — UAMS; Elias Anaissie, MD, Principal Investigator — UAMS; Gal Shafirstein, PhD, Principal Investigator — UAMS